CLINICAL TRIAL: NCT04602780
Title: Evaluating the Revised Work Rehabilitation Questionnaire in Cochlear Implant Users
Brief Title: Evaluating the Revised WORQ in CI Users
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Collaborators: World Hearing Centre (Unknown); Hospital Universitario La Paz (Other); Fiona Stanley Hospital (Other); Wuerzburg University Hospital (Other)
Responsible Party: Principal Investigator, Griet Mertens, Prof., University Hospital, Antwerp
Other Study IDs: 20/23/300
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Hearing Loss
Keywords: Work Rehabilitation Questionnaire; International Classification of Functioning, Disability and Health; Cochlear Implantation
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CI users

SUMMARY:
The Work Related Questionnaire (WORQ) is a 59-item questionnaire of which each item represents an International Classification of Functioning and disability category. The WORQ was modified and reduced to include only questions relevant to Cochlear Implant (CI) users. In this analysis, a multicentre retrospective review of the revised WORQ in CI users was performed, with the revised WORQ as part of the questionnaires used in the regular clinical follow-up of CI users. Experienced CI users' responses on the questions will be evaluated to define the qualifiers for the revised WORQ.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 years
* Adults must wear a MED-EL cochlear implant
* Adults may have the following hearing indications and device fitting:

  * Unilateral cochlear implant with severe-to-profound hearing loss
  * Bilateral cochlear implant with severe-to-profound hearing loss
  * Single sided deafness (SSD) where the poorer ear PTA ≥70 dB HL and the better ear PTA ≤30 dB HL with an interaural threshold gap of ≥40 dB HL.
  * Asymmetrical hearing loss using a cochlear implant in the poorer ear and a hearing aid in the better ear (also known as bimodal fitting). The poorer ear PTA ≥70 dB HL and the better ear PTA >30 dB HL and ≤55 dB HL with an interaural threshold gap of ≥15 dB HL.
* Adults should have a minimum of one year's device experience

Exclusion Criteria

No extra exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Experienced adult CI users
Sampling Method: Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-07-13 (Actual); Study Completion 2020-07-13 (Actual)

PRIMARY OUTCOMES:
Completion of the WORQ questionnaire | One test interval, at least one year after Cochlear Implantation
  Part 1: Work situation and educational background of participants
  * School education
  * Remunerative employment
  Part 2: Daily life functioning of participants
  * Emotional functions
  * Vestibular functions
  * Carrying out daily routine
  * Stress
  * Conversation
  * Communication devices and techniques
  * Tinnitus and dizziness
  * Community life
  * Family relationships
  Part I addresses demographics and relevant background information. In Part 2, participants have to rate to what extent they had problems with a certain task or activity in the last week based on a numerical scale ranging from 0 (no problem) to 10 (complete problem).
  Each individual WORQ item is linked to an ICF qualifier, which is a numerical code that specifies the extent or magnitude of functioning or disability in that ICF category or the extent to which a contextual factor is a facilitator or barrier.

CONTACTS AND LOCATIONS:
Locations (5):
- Fiona Stanley Fremantle Hospital Group, Perth, Australia
- University Hospital Antwerp, Edegem, Belgium
- University Clinic of Würzburg, Würzburg, Germany
- World Hearing Centre, Kajetany, Poland
- Hospital La Paz, Madrid, Spain